CLINICAL TRIAL: NCT04787718
Title: Roles of Almonds in Physical Performance
Brief Title: Almond for Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Mark Kern, Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 59997A
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Muscle Soreness; Energy
MeSH Terms: conditions — Myalgia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond (Experimental): Participants will consume 2.0 oz of raw, shelled, unsalted almonds.
  Interventions: Other: Almond
- Control group (Active Comparator): an isocaloric (2.0 oz raw almonds) amount of unsalted pretzels daily.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Almond — 2.0 oz of raw, shelled, unsalted almonds
  Arms: Almond
Other: Control group — an isocaloric amount of unsalted pretzels
  Arms: Control group

SUMMARY:
Investigators specific aims are to compare the effects of consuming daily snacks of raw, shelled, unsalted almonds (2.0 ounces) versus an isocaloric amount of another commonly consumed snack food (pretzels) on energy (vigor) perception and physical activity, exercise performance (VO2max and measures of strength), strength and power performance as well as muscle soreness recovery after strenuous eccentrically-biased exercise.

DETAILED DESCRIPTION:
To accomplish these aims, investigators will examine whether regular consumption of almonds versus a common snack food over a period of 8 weeks impacts longer term metabolic, physiological and behavioral responses related to energy sensations and exercise capacity/performance.

ELIGIBILITY:
Inclusion Criteria:

* 30-50 years old
* BMI of 23-30

Exclusion Criteria:

* smoking,
* medications known to impact inflammation,
* musculoskeletal limitations and
* use of supplements within 1 month of participation that are known to impact antioxidant
* use of supplements within 1 month of participation that are known to impact inflammatory status

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in energy (vigor) perception | At baseline , at 8 weeks
  Energy (vigor) perception will be assessed using POMS questionnaire
Changes from baseline in exercise performance | At baseline , at 8 weeks
  VO2max will be assessed for measuring exercise performance

SECONDARY OUTCOMES:
Changes from baseline in strength and power performance | At baseline, at 8 weeks
  strength and power performance by be measure by biodex
Changes from baseline in muscle soreness | At baseline, at 8 weeks
  muscle soreness will be measured by DOMES questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Derived] Rayo VU, Cervantes M, Hong MY, Hooshmand S, Jason N, Liu C, North E, Okamoto L, Storm S, Witard OC, Kern M. Almond Consumption Modestly Improves Pain Ratings, Muscle Force Production, and Biochemical Markers of Muscle Damage Following Downhill Running in Mildly Overweight, Middle-Aged Adults: A Randomized, Crossover Trial. Curr Dev Nutr. 2024 Aug 7;8(9):104432. doi: 10.1016/j.cdnut.2024.104432. eCollection 2024 Sep. PMID 39257478